CLINICAL TRIAL: NCT02010840
Title: The Effect of a Father Inclusive Psychoeducation Program on Postnatal Depression: a Randomized Controlled Trial
Brief Title: The Effect of a Father Inclusive Psychoeducation Program on Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Education Bureau, The Government of the Hong Kong Special Administrative Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 748113
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2017-06

CONDITIONS: Pregnancy
Keywords: Depressive symptoms, marital relationship, quality of life
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Psychodeucation program (Experimental): Both couples receive the father inclusive psychoeducation program which consists of a single 3-hour session during pregnancy and two telephone follow up at postpartum.
  Interventions: Behavioral: Psychoeducation program
- Mother only (Active Comparator): Only the women receives the psychoeducation program.
  Interventions: Behavioral: Psychoeducation program
- Control group (No Intervention): Receives usual perinatal care services only

INTERVENTIONS:
Behavioral: Psychoeducation program
  Arms: Mother only; Psychodeucation program

SUMMARY:
Study hypothesis: Childbearing couples who receive the father inclusive psychoeducation program will have: (a) a lower level of depressive symptoms, (b) a higher level of marital relationship, and (c) a higher level of quality of life at 6 weeks, 6 months and one year postpartum than those who receive the usual perinatal care.

DETAILED DESCRIPTION:
Background: Having a first child is a key marker of the transition into parenthood that requires substantial adjustment of couples' life. A recent meta-analysis published in the Journal of American Medical Association reports that both women (23.8%) and men (10.4%) suffer from perinatal depression [1]. The father's involvement during pregnancy can positively influence health outcomes not only for the man, but his partner, and their children [1,2]. However, the effectiveness of father's involvement in prenatal care in preventing paternal and maternal depression, is still unknown.

Aims: This study seeks to: (1) evaluate the effect of a father inclusive psychoeducation program for first-time Chinese mothers and fathers on depressive symptoms (primary outcome), marital relationships and quality of life at 6 weeks, 6 months and one year postpartum; and (2) explore fathers' involvement, their perceived benefits of participating in the program and factors influencing the effectiveness of the program.

Methods: This study employs a longitudinal, randomized, pre and post-test design. A convenience sample of 576 couples will be recruited at antenatal clinics and randomly assigned to one of three groups: (1) the experimental group with both couples receives the intervention on top of usual perinatal care; (2) the comparison group with only the women receives the intervention on top of usual perinatal care; and (3) the control group receives usual perinatal care only. The intervention consists of a single 3-hour session during pregnancy and two telephone follow-up at postpartum week one and week two. Primary outcome on postnatal depression will be assessed by Edinburgh Postnatal Depression Scale. Secondary outcomes on marital relationship and quality of life will be assessed by Dyadic Adjustment Scale and Medical Outcomes Study Short Form 12-item Health Survey, respectively, at baseline, 6 weeks, 6 months and one year postpartum. Process evaluation will be conducted at 6 weeks postpartum using individual telephone interview on 20 couples randomly selected from the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above;
* first-time parents;
* able to speak and read the Chinese language; and
* Hong Kong residents.

Exclusion Criteria:

* couples with past or family psychiatric history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wan Ngai, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychodeucation program: Both couples receive the father inclusive psychoeducation program which consists of a single 3-hour session during pregnancy and two telephone follow up at postpartum.
  Psychoeducation program
- Mother only: Only the women receives the psychoeducation program.
  Psychoeducation program
Period: Overall Study
Arm/Group | Psychodeucation program | Mother only | Control group
Started | 134 | 124 | 130
Completed | 134 | 124 | 130
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychodeucation Program | Mother Only | Control Group | Total
Number analyzed (Participants) | 134 | 124 | 130 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (4) | 32 (4) | 31 (4) | 32 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 65 | 194
  Male | 67 | 62 | 65 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 134 | 124 | 130 | 388

OUTCOME MEASURES:

1. Primary Outcome: Edinburgh Postnatal Depression Scale
Description: Edinburgh Postnatal Depression Scale
Time Frame: 6 weeks postpartum
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Psychodeucation program | Mother only | Control group
Number analyzed (Participants) | 134 | 124 | 130
score on a scale | 41 (0) | 35 (0) | 37 (0)

2. Secondary Outcome: Edinburgh Postnatal Depression Scale
Time Frame: 6 months postpartum
Reporting Status: Not Posted

3. Secondary Outcome: Edinburgh Postnatal Depression Scale
Time Frame: 12 months postpartum
Reporting Status: Not Posted

4. Secondary Outcome: Dyadic Adjustment Scale
Time Frame: 6 weeks postpartum
Reporting Status: Not Posted

5. Secondary Outcome: Dyadic Adjustment Scale
Time Frame: 6 months postpartum
Reporting Status: Not Posted

6. Secondary Outcome: Dyadic Adjustment Scale
Time Frame: 12 months postpartum
Reporting Status: Not Posted

7. Secondary Outcome: Medical Outcomes Study Short Form 12-item Health Survey
Time Frame: 6 weeks postpartum
Reporting Status: Not Posted

8. Secondary Outcome: Medical Outcomes Study Short Form 12-item Health Survey
Time Frame: 6 months postpartum
Reporting Status: Not Posted

9. Secondary Outcome: Medical Outcomes Study Short Form 12-item Health Survey
Time Frame: 12 months postpartum
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The delivery of a psychoeducation programme probably will not lead to serious adverse events, all-caused mortality or other risks.
Arm/Group | Psychodeucation program | Mother only | Control group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT02010840/Prot_SAP_000.pdf